CLINICAL TRIAL: NCT04887636
Title: Baseline Study of Vaginal Microbiota in Healthy Chinses Female Population
Acronym: BSOVM
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-2902
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Vagina Disease; Vaginal Community State Type
Keywords: Vaginal microbiota; Nugent score; Artificial intelligence; Next generation sequencing
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The vaginal secretions were stained with Gram for morphological analysis. The metagenomics or 16s rRNA high-throughput sequencing combined with bioinformatics were used to calculate the structure of the vaginal microbiome flora of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal women group: I. Women of childbearing age who are physically and mentally healthy, have regular menstruation and are between 20-45 years old; II. Women who are evaluated as normal by vaginal microbiome morphological characterization; III. Women who agree to participate in this study and have signed an informed consent form; IV. Those who have full capacity for civil and legal conduct; V. The quality of vaginal samples meets the evaluation requirements of this program.

INTERVENTIONS:
Other:

SUMMARY:
The reproductive tract microecology is an important part of the human microbial system. Microorganisms and the host reproductive tract environment form a stable symbiotic relationship. When pathogens invade or microecology imbalance，it can lead to serious reproductive tract infection.Reproductive tract infection is one of the most common disease among women，and it is a global social and public health problem. Reproductive tract infection is characterized by high morbidity, low cure rate and high recurrence rate.Data from the studies shows that 40% of Chinese women suffer from reproductive tract infections of varying degrees, that is, at least 200 million. Long-term chronic infections can lead to serious consequences such as infertility, tumor, abortion and premature birth. At present, the diagnostic classification of reproductive tract infection is mainly divided into Aerobic vaginitis（AV), Bacterial vaginosis（BV), Vulvovaginal candidiasis（VVC) and Trichomonas vaginitis（TV). The reproductive tract microbiota is complex, but the clinical classification is relatively simple, which makes the treatment lack of precision. More precise treatment，permanent cure and reducing the recurrence rate are the top priorities in the field of medical and health.

DETAILED DESCRIPTION:
At present, the treatment of vaginitis is dominated by anti-pathogen medicine. While killing pathogenic microorganisms, it also inhibits the growth of normal vaginal lactobacillus, which further aggravates the vaginal microecological imbalance and makes it the root of refractory, drug-resistant and recurrent reproductive tract infections.

A growing number of studies show that the key point of the treatment for reproductive tract infections is to adjust the proportion of vaginal microorganism composition, in order to achieve the initial Lactobacillus dominant state, and maintaining the balance of vaginal microecology .

The composition and proportion of microorganisms in the lower reproductive tract influenced by a variety of factors, such as changes in sex hormone levels and phases of the menstrual cycle, sexual activity, antibiotic treatment and use of oral contraceptives, vaginal irrigation, menopause, pregnancy, breastfeeding, diabetes and stress . Also, there are obvious differences between different ethnicities and regions . Therefore, we need to conduct correlation analysis on the microbiota structure and various indicators of the Chinese population, and develop a more reasonable method for classifying lower reproductive tract infections and treatments. According to this classification method, accurate diagnosis of vaginal disease is further carried out, more rational treatment options can be implemented，and the health of patients is effectively improved.

Based on the above background, the study collected DNA from vaginal secretions from about 10,000 healthy Chinese women of reproductive age. And the DNA was tested by next genetic sequencing.The data obtained in this project will establish the baseline of the lower reproductive tract microbiome of Chinese population, and will be used for future research and comparison. The results will be used to explore the comparison of the lower reproductive tract flora of the population in different regions of China, and of the Chinese population with other ethnicities worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age who are physically and mentally healthy, have regular menstruation and are between 20-45 years old;
* Women who are evaluated as normal by vaginal microbiome morphological characterization;
* Women who agree to participate in this study and have signed an informed consent form;
* Those who have full capacity for civil and legal conduct;
* The quality of vaginal samples meets the evaluation requirements of this program.

Exclusion Criteria:

* The sampling quality of vaginal secretions does not meet the research study requirements;
* The quality or format of the slide collection of vaginal smears does not meet the requirements;
* Women with severe physical or mental illness;
* Users of hormone therapy and antibiotic drugs;
* Women with insufficient compliance with this study;
* Women who are participating in other coinciding clinical drug or medical device trials.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of childbearing age who are physically and mentally healthy, have regular menstruation and are between 20-45 years old;
Study Population: The comparison of the lower reproductive tract flora of the population in different regions of China, and of the Chinese population with other ethnicities worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Nugent score | 1 year
  The morphological manifestations of vaginal microflora were observed by the examiner under the microscope, and the vaginal microecological results were evaluated according to the Nugent score.Nugent Scoring System（0-10）for Gram-Stained Vaginal Smears Total Score：0-3 Normal； 4-6 Intermediate；7-10 Bacterial Vaginosis
Next generation sequencing | 1 year
  16s rRNA gene sequencing and metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ma B, Forney LJ, Ravel J. Vaginal microbiome: rethinking health and disease. Annu Rev Microbiol. 2012;66:371-89. doi: 10.1146/annurev-micro-092611-150157. Epub 2012 Jun 28. PMID 22746335
- [Background] Knight R, Callewaert C, Marotz C, Hyde ER, Debelius JW, McDonald D, Sogin ML. The Microbiome and Human Biology. Annu Rev Genomics Hum Genet. 2017 Aug 31;18:65-86. doi: 10.1146/annurev-genom-083115-022438. Epub 2017 Mar 20. PMID 28375652
- [Background] White BA, Creedon DJ, Nelson KE, Wilson BA. The vaginal microbiome in health and disease. Trends Endocrinol Metab. 2011 Oct;22(10):389-93. doi: 10.1016/j.tem.2011.06.001. Epub 2011 Jul 13. PMID 21757370
- [Background] Srinivasan S, Liu C, Mitchell CM, Fiedler TL, Thomas KK, Agnew KJ, Marrazzo JM, Fredricks DN. Temporal variability of human vaginal bacteria and relationship with bacterial vaginosis. PLoS One. 2010 Apr 15;5(4):e10197. doi: 10.1371/journal.pone.0010197. PMID 20419168
- [Background] Crucitti T, Hardy L, van de Wijgert J, Agaba S, Buyze J, Kestelyn E, Delvaux T, Mwambarangwe L, De Baetselier I, Jespers V; Ring Plus study group. Contraceptive rings promote vaginal lactobacilli in a high bacterial vaginosis prevalence population: A randomised, open-label longitudinal study in Rwandan women. PLoS One. 2018 Jul 23;13(7):e0201003. doi: 10.1371/journal.pone.0201003. eCollection 2018. PMID 30036385
- [Background] Riggs M, Klebanoff M, Nansel T, Zhang J, Schwebke J, Andrews W. Longitudinal association between hormonal contraceptives and bacterial vaginosis in women of reproductive age. Sex Transm Dis. 2007 Dec;34(12):954-9. PMID 18077845
- [Background] Sobel JD, Kaur N, Woznicki NA, Boikov D, Aguin T, Gill G, Akins RA. Conventional oral and secondary high dose vaginal metronidazole therapy for recurrent bacterial vaginosis: clinical outcomes, impacts of sex and menses. Infect Drug Resist. 2019 Jul 24;12:2297-2307. doi: 10.2147/IDR.S213853. eCollection 2019. PMID 31413606
- [Background] Ravel J, Gajer P, Abdo Z, Schneider GM, Koenig SS, McCulle SL, Karlebach S, Gorle R, Russell J, Tacket CO, Brotman RM, Davis CC, Ault K, Peralta L, Forney LJ. Vaginal microbiome of reproductive-age women. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4680-7. doi: 10.1073/pnas.1002611107. Epub 2010 Jun 3. PMID 20534435
- [Background] France MT, Ma B, Gajer P, Brown S, Humphrys MS, Holm JB, Waetjen LE, Brotman RM, Ravel J. VALENCIA: a nearest centroid classification method for vaginal microbial communities based on composition. Microbiome. 2020 Nov 23;8(1):166. doi: 10.1186/s40168-020-00934-6. PMID 33228810
- [Background] Mizock BA. Probiotics. Dis Mon. 2015 Jul;61(7):259-90. doi: 10.1016/j.disamonth.2015.03.011. Epub 2015 Apr 25. No abstract available. PMID 25921792
- [Background] Tao Zhi, Liao Qinping. Research progress and clinical significance of vaginal microecology. Journal of Practical Obstetrics and Gynecology, 2018, 34(10):721-723.
- [Background] Qin-ping Liao, Dai Zhang. Current status and research progress of diagnosis and treatment of female reproductive tract infections in China. International Journal of Obstetrics and Gynecology, 2011(06):8-10